CLINICAL TRIAL: NCT01718093
Title: A Pilot Study to Assess the Glucose Lowering Effect of Metformin and Sitagliptin in Adolescents With Type 1 Diabetes Mellitus
Brief Title: A Pilot Study to Assess the Glucose Lowering Effect of Metformin and Sitagliptin in Adolescents With Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Luisa M. Rodriguez, Assistant Professor - Department of Pediatrics - Endocrinology and Metabolism, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-29924; DK096067 (Other: NIH)
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Type 1 Diabetes
Keywords: Adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Insulin plus sitagliptin (Active Comparator): The subjects continued their usual insulin regimen throughout the study. Sitagliptin was started and continued at 50 mg orally twice daily
  Interventions: Drug: Sitagliptin
- Insulin plus metformin (Active Comparator): The subjects continued their usual insulin regimen throughout the study. Metformin was started at 500 mg orally daily. The dose was increased over a 2 week period up to 2,000 mg per day as tolerated.
  Interventions: Drug: Metformin
- Insulin plus sitagliptin and metformin (Active Comparator): The subjects continued their usual insulin regimen throughout the study. Sitagliptin was started and continued at 50 mg orally twice daily. Metformin was started at 500 mg orally daily. The dose was increased over a 2 week period up to 2,000 mg per day as tolerated.
  Interventions: Drug: Sitagliptin + Metformin

INTERVENTIONS:
Drug: Sitagliptin — up to 50 mg twice a day
  Other Names: Januvia
  Arms: Insulin plus sitagliptin
Drug: Metformin — up to 1000 mg twice a day
  Other Names: Glucophage
  Arms: Insulin plus metformin
Drug: Sitagliptin + Metformin — up to 50/1000 mg twice a day
  Other Names: Sitagliptin + Metformin = Janumet
  Arms: Insulin plus sitagliptin and metformin

SUMMARY:
The purpose of this study is to see if the use of metformin and sitagliptin used in conjunction with insulin can improve the blood sugars of teenagers with Type 1 diabetes.

DETAILED DESCRIPTION:
* The study will include a total of 4 visits. The time period between the very first visit and the very last visit will be between 10 and 15 weeks. Each participant will be randomized to one of the 3 groups in the study. The groups are as follows:
* Group 1: Insulin and sitagliptin
* Group 2: Insulin and metformin
* Group 3: Insulin and combination of sitagliptin and metformin
* The study is a randomized open label design. All subjects will undergo a screening visit; if inclusion and exclusion criteria are fulfilled they will be enrolled in the study. At the time of enrollment the subject will continue their home insulin regimen and will be randomized to an add an oral hypoglycemic agent(s) : metformin, sitagliptin or combination therapy (metformin and sitagliptin). The total duration on study medication will be 6 weeks. All subjects will undergo a baseline mixed meal tolerance test (MMTT) in their standard or usual insulin Each subject will undergo a total of two studies. Blood draws will be necessary.

ELIGIBILITY:
Inclusion Criteria:

* Age of 13 to 18 years
* HbA1c >7.5% but <10%
* Subjects must be on intensive insulin management
* Tanner stage greater than or equal to 4
* Must have T1DM for at least one year , T1DM defined by ADA criteria and having at least one of the following antibodies: Anti-GAD, Anti-islet, Anti-insulin
* C-peptide > 0.6 ng/ml

Exclusion Criteria:

* Type 2 diabetes
* History of any other chronic condition (except hypothyroidism stable on medications)
* Actively taking medications that may affect glucose excursions (steroids or oral contraceptives)
* Evidence of anemia, clinically significant elevation of the liver enzymes (3 X normal), amylase or lipase (2 X normal), abnormal triclycerides (3 X normal), abnormal renal function test
* An unsupportive family environment and pregnant or lactating females

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To determine the glucose lowering effect of metformin and sitagliptin alone and as combination therapy when used as adjuncts to insulin in adolescents with T1DM. | 10 - 15 weeks
  Glucose concentrations and AUC glucose calculation

CONTACTS AND LOCATIONS:
Overall Officials: Luisa M. Rodriguez, MD, MS, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No